CLINICAL TRIAL: NCT05919862
Title: Three-dimensional Positional Accuracy of Dental Implant Placement Using a Haptic and Machine Vision Controlled Collaborative Surgery Robot: a Pilot Randomized Controlled Trial
Brief Title: Accuracy of Dental Implant Placement Using a Collaborative Surgery Robot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Maurizio Tonetti, Professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SH9H-2023-05
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Dental Implant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot system (Experimental): Prosthetically guided Implant placement utilising robotic surgery based on a digital plan.
  Interventions: Procedure: Robot system
- Freehand surgery (Sham Comparator): Freehand implant placement by experienced surgeon.
  Interventions: Procedure: Freehand surgery

INTERVENTIONS:
Procedure: Robot system — Prosthetically guided Implant placement utilising robotic surgery based on a digital plan
  Arms: Robot system
Procedure: Freehand surgery — Freehand implant placement by experienced surgeon.
  Arms: Freehand surgery

SUMMARY:
For free hand dental implant placement, a key difficulty is to accurately control the position. Improving precision of dental implant placement is considered important for safety and efficacy of tooth replacement with dental implants. The goal of this randomized controlled trial is to compare the positional implant accuracy, and patient reported outcomes comparing two methods of implant placement: the use of a robotic assisted surgery and freehand surgery. Patients requiring single tooth replacement with a dental implant will be digitally planned using a CBCT and an intraoral digital scan. Subjects will be randomized to one of the two treatment modalities based on the plan. The accuracy of placement will be assessed evaluating the difference between the planned and the actual position using a CBCT immediately after surgery. Subjects will be followed up for one year to assess both patient reported and professional outcomes.

DETAILED DESCRIPTION:
For free hand dental implant placement, a key difficulty is to accurately control the position. Improving precision of dental implant placement is considered important for safety and efficacy of tooth replacement with dental implants. In particular, more precise implant placement is expected to yield a better restoration both in terms of aesthetics and ability for self-performed oral hygiene and thus prevention of peri-implant diseases. The goal of this randomized controlled trial is to compare the positional implant accuracy, and patient reported outcomes comparing two methods of implant placement: the use of a robotic assisted surgery and freehand surgery. Patients requiring single tooth replacement with a dental implant will be digitally planned using a CBCT and an intraoral digital scan. Subjects will be randomized to one of the two treatment modalities based on the plan. The accuracy of placement will be assessed evaluating the difference between the planned and the actual position using a CBCT immediately after surgery. Subjects will be followed up for one year to assess both patient reported and professional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a single missing tooth to be replaced with a dental implant
* With sufficient bone volume and keratinized tissue at edentulous site
* Willing to comply with research appointments/schedule.

Exclusion Criteria:

* Pregnancy or intention to become pregnant at any point during the study duration
* With any systemic diseases/conditions that are contraindications to dental implant treatment
* Inability or unwillingness of individual to give written informed consent
* Inability of follow-up according to the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Implant positional accuracy | Immediately after surgery
  Implant accuracy will be measured as distance discrepancy at implant platform and implant apex, and angular discrepancy of implant axis between the digital plan and the actual position of the implant assessed digitally at the end of the procedure. Pre- and post-operative CBCT will be used for measurement.
Peri-implant soft tissue health | 12 month follow-up
  Bleeding on probing and probing depth will be recorded, by probing gently around implant-supported restoration at six points: mesial-buccal, mid-buccal, distal-buccal, mesial-lingual, mid-lingual, and distal-lingual, using UNC-15 periodontal probe. This is defined according to the peri-implant health case definition by Berglundh et al 2017 and the ID-COSM international consensus conference

SECONDARY OUTCOMES:
Local integrity of the alveolar bone | Immediately after surgery
  The thickness of the buccal and lingual bone plates 1, 3, and 5 mm apical to the implant platform on post-surgery CBCT
Discomfort perception | During surgery
  Patient discomfort perception during surgery will be recorded using visual analogue scale (VAS with range from 0 to 10 with 10 being the highest possible pain experience)
Pain perception | immediately after surgery, and 1 to 7 days after surgery
  Patient pain perception after surgery will be recorded using visual analogue scale (VAS with range from 0 to 10 with 10 being the highest possible pain experience) .
Esthetics of the restoration | 12-months follow-up after delivery of crown
  Assessed using the PES-WES scale as reported by Belser et al.with the scale ranging from 0 to 14 (worst to best)
Cytokine concentrations in PISF | 12-months follow-up after delivery of crown
  Cytokine concentration in peri-implant sulcus fluid assesed by MULTIPLEX ELISA as concentrations of IL-1, TNF, IL-6 with lower concentrations reflecting less local inflammation
Submarginal microbiome | 12-months follow-up after delivery of crown
  16S assessment of microbiome diversity (Shannon index) with greater diversity representing a more stable microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Tonetti Maurizio, PhD, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Department of Oral and Maxillofacial Implantology, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No